CLINICAL TRIAL: NCT06061666
Title: TILIA for inSomnia During HOrmonal Therapy in Breast Cancer Survivors
Brief Title: Treatment of Insomnia in Patients With Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5175
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Insomnia
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (Experimental): Group treated with MG-C of Tilia tomentosa
  Interventions: Other: Tilia tomentosa Concentrated - Glycerine macerate (C-GM) vs Placebo (1 gtt/10 kg/day before bedtime for 15 days)
- Placebo Group (Placebo Comparator): Group treated with placebo
  Interventions: Other: Tilia tomentosa Concentrated - Glycerine macerate (C-GM) vs Placebo (1 gtt/10 kg/day before bedtime for 15 days)

INTERVENTIONS:
Other: Tilia tomentosa Concentrated - Glycerine macerate (C-GM) vs Placebo (1 gtt/10 kg/day before bedtime for 15 days) — Self-administration of the food supplement or placebo (1 gtt/10 kg/day before bedtime for 15 days)

SUMMARY:
Insomnia, defined as difficulty falling asleep, staying asleep, or waking up too early at least three times a week for at least 3 months, (American Psychiatric Association 2013) is a common disorder both in the general population and in cancer patients, but it is particularly common in breast cancer patients. (Davidson JR, 2002) (Savard J, 2001). Unfortunately, this issue is often not recognized and is not adequately addressed in common clinical practice (Zhou ES, 2017). Emotional distress, stress after surgery, and side effects of cancer treatments, particularly those related to hormone therapy, all contribute to the onset of insomnia, which, in turn, can contribute to a poor quality of life, to greater fatigue in carrying out daily life activities, to worsening physical and emotional discomfort (Kyle SD, 2010) (Bolge SC, 2009) (Sarsour K, 2011).

To date, insomnia in common clinical practice is an often overlooked problem. Patients report that healthcare providers rarely pay attention to sleep disorders and even if they are evaluated, treatment recommendations tend to focus primarily on prescribing medications (Siefert ML, 2014).

Gemmotherapy is a young branch of phytotherapy developed in the second half of the last century. This branch bases its principles on the therapeutic potential of the meristematic tissues of plants and uses products called glycerine macerates (GM) obtained according to the method of cold maceration of meristematic tissues in water, alcohol and glycerol created by Dr. Pol Henry in the last century or according to the Pharmacopoeias.

The use of concentrated GM (C-GM) has spread (Andrianne, 2008 and 2012). These C-MGs are approximately 10 times more concentrated than traditional GMs, and are therefore traditionally used at lower doses (adults: approximately 5-15 gtt/day) than those used for diluted extracts (adults: up to 1 gtt/kg/day ).

Tilia tomentosa, whose fresh buds are used, is traditionally indicated in all cases of insomnia in adults and children. Its action is carried out by inducing sleep and increasing its duration. In phytotherapy it is recommended in neuroses but also as an antispasmodic, in heart palpitations and in spasmophilia. No type of acute or chronic toxicity is known for this C-GM.

In the proposed study we want to evaluate the action of C-GM from Tilia tomentosa, extracted according to the Pharmacopoeias, for the treatment of insomnia in patients with breast cancer on hormone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients capable of giving informed consent
* Patients undergoing surgery to remove breast tumors and undergoing hormone therapy (any stage)
* Patients who present a score > 5 on the "Pittsburgh Sleep Quality Index (PSQI)" questionnaire on sleep quality
* Patients aged between 18 and 65 years

Exclusion Criteria:

* Children under 18 and people over 65
* Pregnant or breastfeeding women
* Patients with breast cancer undergoing chemotherapy and/or radiotherapy
* Serious concomitant diseases (other neoplasms, liver failure, renal failure, and hyperthyroidism, ulcerative colitis, Crohn's disease)
* Patients being treated with antibiotics in the month preceding screening
* Patients being treated with drugs that alter the sleep-wake rhythm (anxiolytics, hypnotics, non-benzodiazepine hypnotics, major sedatives, antipsychotics, antiepileptics, opiates)
* Known hypersensitivity to Tilia tomentosa

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Tilia tomentosa glyceric macerate effectiveness against insomnia of brest cancer patients | T1: 15 days, and T2: 75 days
  evaluate the effect of the Tilia tomentosa C-GM food supplement in contributing to the physiological restoration of the quality and duration of sleep in patients undergoing breast cancer surgery and hormone therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di Scienze di Laboratorio e Infettivologiche, Rome, Italy